CLINICAL TRIAL: NCT05408455
Title: Effect of Expiratory Muscle Training in Bronchiectasis Patients
Brief Title: Expiratory Muscle Training in Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ayşenur Yılmaz, MSc Pt, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 646873
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; cough strength; expiratory muscle training; exercise capacity
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMST (Expiratory Muscle Streght Training) group (Experimental): EMST at a pressure value between 50-75% will be applied for 8 weeks, 3 days a week and 24 sessions in total.
  Interventions: Other: EMST150 (Expiratory muscle training)
- Sham EMST Group (Sham Comparator): EMST without threshold loading will be applied for 8 weeks, 3 days a week and 24 sessions in total.
  Interventions: Other: Sham EMST150 (Expiratory muscle training)

INTERVENTIONS:
Other: EMST150 (Expiratory muscle training) — Respiratory exercise device (Expiratory muscle trainer) developed for the expiratory muscles, and resistant expiratory muscle training were applied. Threshold loading was applied to the cases at approximately 30% of the respiratory muscle strength values measured in the 1st week. In respiratory muscle training, the pressure value was increased according to the tolerance of the patient and training was given at a pressure value between 50-75%. The subjects were asked to do 10 vigorous expirations at the adjusted pressure value by doing normal inspiration for expiratory muscle training in a comfortable sitting position. This program was applied in 3 sets in the same way for approximately 30 minutes. It was continued 3 days a week for 8 weeks
  Arms: EMST (Expiratory Muscle Streght Training) group
Other: Sham EMST150 (Expiratory muscle training) — The subjects were asked to perform normal inspiration and then exhale 10 times for expiratory muscle training without threshold loading. This program was applied in 3 sets in the same way for approximately 30 minutes. It will continue 3 days a week for 8 weeks
  Arms: Sham EMST Group

SUMMARY:
Reduced exercise tolerance is commonly reported in patients with bronchiectasis. The purpose of this study is to evaluate the effects of expiratory muscle training (EMT) and sham EMT (control) on exercise capacity, respiratory function and respiratory muscle strength, cough strength and health related quality of life in patients with bronchiectasis.

DETAILED DESCRIPTION:
Disruption of the mucociliary clearance mechanism in patients with bronchiectasis leaves the lungs vulnerable. With the accumulation of secretions, a vicious cycle of bacterial infection and inflammation begins. Intense inflammation causes damage and bronchial wall weakness. Problems arise with effective coughing. This leads to decreased clearance of secretions, resulting in decreased expiratory flow. Symptoms of bronchiectasis; often productive cough, dyspnea, fatigue and wheezing. Altered pulmonary mechanics, inadequate gas exchange, decreased muscle mass, and accompanying psychological problems can cause dyspnea and decreased exercise capacity, thus reducing quality of life. Exercise capacity may also decrease in individuals with bronchiectasis due to increased dyspnea perception and limitation of expiratory flow. The need for safe and viable exercise interventions to reduce the burden of the disease is evident in individuals with bronchiectasis. Respiratory muscle training is applied by using skeletal muscle training principles in order to increase respiratory muscle strength and endurance, to correct the length-tension relationship of respiratory muscles and to increase respiratory capacity. Decreased expiratory muscle strength is associated with decreased quality of life and exercise tolerance. In addition, in a study, it was shown that in addition to expiratory muscle weakness, expiratory muscle endurance decreases in respiratory patients. This decrease is closely related to the severity of airway obstruction and the decrease in the strength of other muscle groups.

In order to meet the increased metabolic needs during exercise and to keep gas exchange at a sufficient level, patients with bronchiectasis; they must increase minute ventilation as appropriate. These patients with expiratory flow limitation at rest breathe at higher lung volumes to increase ventilation during exercise, and as a result, adverse conditions such as worsening of dynamic hyperinflation, increased intrinsic PEEP, increased workload on respiratory muscles and dyspnea are observed. As a result, these patients cannot achieve high levels of tidal volume and ventilation. In addition, significantly reduced maximal voluntary ventilation in patients with flow-limited bronchiectasis; It is also related to airway obstruction and mechanical deterioration. Decreased exercise capacity has also been shown to be associated with peak exercise desaturation. Those with abnormal lung mechanics (low FEV1, FVC, and tidal expiratory flow limitation) and high dyspnea score measured by MRC reflect a decrease in exercise capacity. In a study in bronchiectasis, maximal inspiratory and maximal expiratory respiratory muscle strengths evaluated with an intraoral pressure measurement device had similar demographic characteristics. significantly lower than in healthy individuals. However, in the respiratory muscle trainings, inspiratory muscle training was emphasized and expiratory muscle training was never given.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients who do not meet the definition of exacerbation,
* Those with a diagnosis of non-CF bronchiectasis,
* Patients are between the ages of 18-70
* Patients without acute and/or chronic respiratory failure,
* Patients who do not have any contraindications for the physiotherapy method to be applied.

Exclusion Criteria:

* Those with a history of pneumothorax,
* Patients younger than 18 years
* Patients older than 70 years
* Presence of cor pulmonale and/or heart failure,
* Patients with hemoptysis,
* Those with a recent history of acute myocardial infarction,
* Presence of spinal cord injury,
* Those with unstable intervertebral disc, rib fracture,
* Patients with severe osteoporosis,
* Those who had an infective exacerbation during the physiotherapy application period,
* Those who are found to have respiratory distress that will require hospitalization,
* If there is a wound in the application area,
* If there is infection or hemorrhage in the application area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-24 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | Baseline to 8 weeks
  Exercise capacity using 6-minute walk test
Cough strength | Baseline to 8 weeks
  Cough strength using PEF meter
Respiratory muscle strength | Baseline to 8 weeks
  Respiratory muscle strength is measured through maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) using cosmed pony fx.

SECONDARY OUTCOMES:
Leicester Cough Questionnaire | Baseline to 8 weeks
  Health related quality of life is assessed with Leicester Cough Questionnaire. The total score range is 3-21 and domain scores range from 1-7; a higher score indicates a better quality of life.
Modified Medical Research Council Dyspnea Scale (MMRC) | Baseline to 8 weeks
  Dyspnea severity is assessed with The Modified Medical Research Council Dyspnea Scale (MMRC).The mMRC scale is a self-rating tool to measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness except on strenuous exercise; 4, too breathless to leave the house, or breathless when dressing or undressing.
Bronchiectasis Severity Index | Baseline to 8 weeks
  Severity of disease is assessed with Bronchiectasis Severity Index. The total score is calculated by summing the scores for each variable and can range from 0 to 26 points. According to the overall score, patients are classified into three classes: patients with low BSI score (0-4 points), intermediate BSI score (5-8 points), high BSI score (≥9 points).
St. George's Respiratory Questionnaire (SGRQ) | Baseline to 8 weeks
  Health related quality of life is assessed with St. George's Respiratory Questionnaire (SGRQ).SGRQ scores range from 0 to 100, with higher scores indicating worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur yılmaz, MSc Pt, Study Director — Pamukkale University; orçin telli atalay, Doç, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No